CLINICAL TRIAL: NCT05568238
Title: Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated Fascial Traction (VAWCPOM) in Patients With Open Abdomen - a Prospective Multi-center Cohort Study
Brief Title: Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated Fascial Traction in Patients With Open Abdomen
Acronym: VAWCPOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Petersson, Principal investigator, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131-22
Record Dates: First submitted 2022-09-10; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Open Abdomen; Temporary Abdominal Closure; Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated fascial traction (Other): Incisional hernia incidence for patients treated with Vacuum Assisted Wound Closure and Permanent On-lay Mesh mediated fascial traction
  Interventions: Procedure: Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated fascial traction (VAWCPOM)

INTERVENTIONS:
Procedure: Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated fascial traction (VAWCPOM) — Vacuum Assisted Wound Closure and Permanent On-lay Mesh-mediated fascial traction (VAWCPOM) in patients with open abdomen.

SUMMARY:
Open abdomen therapy is used in trauma and non-trauma patients where the abdomen is not possible to close, or the intraabdominal conditions is not suitable for closure. In 2007, a new technique that made use of negative pressure wound therapy and mesh-mediated fascial traction for closure of the open abdomen was described from the Department of Surgery in Malmö, Sweden. With this new technique, fascial closure rates were high but long-term incisional hernia formation was seen in approximately half of the patients alive after five years. To overcome the high incisional hernia incidence, a new technique utilizing a permanent on-lay mesh for traction and reinforcement of the incision at fascial closure was developed.

Hypothesis Lower incisional hernia rates in comparison with literature reported results of other techniques for open abdomen treatment, with similar complication rates.

Aims To evaluate early and late clinical outcome of the novel vacuum-assisted wound closure and permanent on-lay mesh-mediated fascial traction technique.

Design A prospective six-center cohort study in Sweden and Denmark. Study inclusion during a two-year period or longer to include at least 100 patients. Statistical analysis will be done by intention-to-treat and as sub-group per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

• All patients ≥18 years old treated with an open abdomen with a midline incision, regardless of indication.

Exclusion Criteria:

* Patient declining participation
* Existing incisional hernia or primary ventral hernia ≥3 cm
* Existing mesh in the abdominal wall, located in the midline and irrespective of mesh size
* Existing ostomy/parastomal hernia located in a position that prevents the VAWCPOM technique to be utilized
* Closure of the abdomen at first dressing change, e. g. without mesh traction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia at 1 year | 1 year, year 1
  Incidence of incisional hernia after open abdomen closure with the technique

SECONDARY OUTCOMES:
Fascial closure rate | During hospital stay
  Percentage of patients possible to closed with the technique
Complications | Up to 12 weeks
  Complications related to the technique
Incisional hernia | Through study completion, 3 years
  Incisional hernia incidence after three years
EQ5D | Through study completion, 3 years
  Patient reported outcome of generic quality of life
HERO | Through study completion, 3 years
  Patient reported outcome of abdominal wall function and discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Pettersson, Ass prof, Principal Investigator — Lund University, Sweden. Department of Surgery Skane university hospital, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersson P, Montgomery A, Petersson U. Vacuum-Assisted Wound Closure and Permanent Onlay Mesh-Mediated Fascial Traction: A Novel Technique for the Prevention of Incisional Hernia after Open Abdomen Therapy Including Results From a Retrospective Case Series. Scand J Surg. 2019 Sep;108(3):216-226. doi: 10.1177/1457496918818979. Epub 2018 Dec 21. PMID 30574843